CLINICAL TRIAL: NCT00763360
Title: To Compare the Ability of DiscoVisc® Ophthalmic Viscosurgical Device (OVD) to Protect the Corneal Endothelium and Maintain Anterior Chamber Space With Healon® and Amvisc® PLUS During Cataract Surgery.
Brief Title: To Compare the Ability of DiscoVisc® OVD to Protect the Corneal Endothelium and Maintain Anterior Chamber Space With Healon® and Amvisc® PLUS During Cataract Surgery.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: AUS-S-07-01
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2012-01-24 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2011-12

CONDITIONS: Cataract
Keywords: Cataract
MeSH Terms: conditions — Cataract | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- DisCoVisc® (Experimental): DisCoVisc® Ophthalmic Viscosurgical Device
  Interventions: Device: DisCoVisc®
- Healon (Active Comparator): Healon
  Interventions: Drug: Healon
- Amvisc Plus (Active Comparator): Amvisc Plus
  Interventions: Drug: Amvisc Plus

INTERVENTIONS:
Device: DisCoVisc® — Injection of DisCoVisc® Ophthalmic Viscosurgical Device (OVD) into the anterior chamber prior to and throughout the cataract surgery procedure
  Arms: DisCoVisc®
Drug: Healon — Injection of Healon into the anterior chamber prior to and throughout the cataract surgery procedure
  Arms: Healon
Drug: Amvisc Plus — Injection of Amvisc Plus into the anterior chamber prior to and throughout the cataract surgery procedure
  Arms: Amvisc Plus

SUMMARY:
The objective of the study is to assess how DisCoVisc Ophthalmic Viscosurgical Device (OVD) compares with Healon and Amvisc Plus in the protection of corneal endothelial cells, and the ability to maintain anterior chamber space, in routine cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to understand and sign a document of informed consent;
* Patients aged ≥49 years with age-related cataract formation;
* Patients planning to undergo surgical removal of cataract by phacoemulsification with implantation of a posterior chamber intraocular lens;
* Patients that have healthy eyes excluding the formation of cataract.

Exclusion Criteria:

* pseudoexfoliation syndrome with glaucoma or zonular compromise in the operative eye;
* A congenital ocular anomaly (e.g., aniridia, congenital cataract) in the operative eye;
* Iris atrophy in the operative eye;
* Glaucoma (including pseudoexfoliation or pigmentary) or any causes of compromised outflow in the operative eye;
* Any abnormality which prevents reliable Goldmann applanation tonometry in the operative eye;
* Ocular hypertension (lntraocular Pressure (IOP) > 21 mmHg) in the operative eye at the baseline exam;
* Corneal abnormality that results in a poor endothelial cell photograph and prevents reliable endothelial cell density measurement;
* Baseline endothelial cell density < 1500 cells/mm2, in the operative eye;
* Planned multiple procedures during cataract/Intraocular Lens (IOL) implantation surgery (e.g., trabeculoplasty, corneal transplant). NOTE: A minor relaxing keratotomy
* Patients 48 years of age or younger;
* Proliferative diabetic retinopathy in the operative eye;
* Uncontrolled diabetes mellitus;
* Marfan's Syndrome;
* An ocular disease and/or condition that may compromise results;
* A history of chronic or recurrent inflammatory eye disease (e.g. iritis, scleritis, uveitis, iridocyclitis, rubeosis iritis) in the operative eye;
* Lens for the correction of astigmatism may be performed;
* Previous ocular trauma to the operative eye (this includes previous intraocular surgery and traumatic cataract). NOTE: history of non-invasive laser surgery (with the exception of laser treatment for PDR) is acceptable for inclusion;
* A non-functional fellow eye;
* Participation in any other clinical study within the 30 days before surgery

Min Age: 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2008-05; Primary Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were undergoing a cataract operation and were recruited from surgery during 2008 to 2010
Pre-assignment Details: Patients were screened prior to cataract operation
Period: Overall Study
Arm/Group | DisCoVisc® | Healon | Amvisc Plus
Started | 61 | 60 | 63
Completed | 61 | 58 | 63
Not Completed | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DisCoVisc® | Healon | Amvisc Plus | Total
Number analyzed (Participants) | 61 | 60 | 63 | 184
Age Continuous [Mean (Standard Deviation); unit: years] | 73.97 (9.03) | 75.56 (7.6) | 75.51 (8.49) | 75.01 (8.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 40 | 43 | 117
  Male | 27 | 20 | 20 | 67

OUTCOME MEASURES:

1. Primary Outcome: Endothelial Cell Count Change From Baseline
Description: Change in endothelial cell count compared to baseline. Endothelial cell count peformed by counting of cells on photographic image of endothelium.
Time Frame: one month
Population: Only those participants that had endothelial cell counts at both baseline and follow-up were included in this analysis.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | DisCoVisc® | Healon | Amvisc Plus
Number analyzed (Participants) | 57 | 58 | 61
Percent change from baseline | -7.91 (16.49) | -5.11 (19.41) | -4.92 (13.89)

2. Primary Outcome: Investigator Reported Space Maintenance
Description: Maintenance of the anterior chamber/dome during cataract surgery. This was rated by the surgeon in one of 4 categories: "Full Chamber Maintained", "Working Space Maintained", "Shallow", "Flat". Space maintenance was reported during Capsulorhexis, Hydrodissection, Phacoemulsification, and IOL insertion.
Time Frame: During surgical procedure
Measure: Number; unit: participants
Arm/Group | DisCoVisc® | Healon | Amvisc Plus
Number analyzed (Participants) | 61 | 58 | 61
participants
  Capsulorhexis - full chamber maintained | 59 | 26 | 61
  Capsulorhexis - working space maintained | 2 | 26 | 1
  Capsulorhexis - shallow | 0 | 5 | 1
  Capsulorhexis - flat | 0 | 1 | 0
  Hydrodissection - full chamber maintained | 52 | 10 | 45
  Hydrodissection - working space maintained | 8 | 22 | 10
  Hydrodissection - shallow | 1 | 16 | 6
  Hydrodissection - flat | 0 | 10 | 2
  Phacoemulsification - full chamber maintained | 59 | 55 | 62
  Phacoemulsification - working space maintained | 2 | 3 | 1
  Phacoemulsification - shallow | 0 | 0 | 0
  Phacoemulsification - flat | 0 | 0 | 0
  IOL insertion - full chamber maintained | 59 | 48 | 63
  IOL insertion - working space maintained | 2 | 8 | 0
  IOL insertion - shallow | 0 | 1 | 0
  IOL insertion - flat | 0 | 1 | 0

3. Secondary Outcome: Change in Corneal Thickness
Description: Change in corneal thickness from baseline, measured in millimeters. Measurement performed by pachymetry.
Time Frame: 1 month
Population: Subjects that did not have both baseline and 1 month values were not included in this analysis.
Measure: Median (Standard Deviation); unit: millimeters
Arm/Group | DisCoVisc® | Healon | Amvisc Plus
Number analyzed (Participants) | 57 | 57 | 61
millimeters | 0.53 (0.04) | 0.54 (0.04) | 0.53 (0.04)

4. Secondary Outcome: Corneal Clarity
Description: Evaluation of corneal clarity as assessed by levels of aqueous flare and aqueous cells. Evaluations were based on the surgeons judgement and graded on a scale. Aqueous flare was graded on the following scale: No visible flare, mild, moderate, severe. Aqueous cells were graded on the following scale: no cells, 1-20 cells, 10-50 cells, too many cells to count, cells frozen.
Time Frame: 2 weeks
Population: Data from subjects for whom this evaluation was not performed is not included in this analysis.
Measure: Number; unit: units on a scale
Arm/Group | DisCoVisc® | Healon | Amvisc Plus
Number analyzed (Participants) | 61 | 58 | 63
units on a scale
  Aqueous flare - no visible flare | 2 | 2 | 1
  Aqueous flare - mild | 53 | 54 | 59
  Aqueous flare - moderate | 6 | 4 | 3
  Aqueous flare - severe | 0 | 0 | 0
  Aqueous cells - no cells | 0 | 0 | 0
  Aqueous cells - 1-10 cells | 10 | 8 | 11
  Aqueous cells - 10-50 cells | 34 | 37 | 37
  Aqueous cells - too many cells to count | 16 | 15 | 15
  Aqueous cells - cells frozen | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Description: All adverse events were recorded by Principal Investigator.
Arm/Group | DisCoVisc® | Healon | Amvisc Plus
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/60 | 0/63
Other Adverse Events (participants affected / at risk) | 0/61 | 0/60 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No